CLINICAL TRIAL: NCT00571688
Title: Does Risperidone Consta Reduce Relapse and Rehospitalization in Bipolar Disorder?
Acronym: Consta
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Vanderbilt University (Other)
Collaborators: Ortho-McNeil Janssen Scientific Affairs, LLC (Industry)
Responsible Party: Principal Investigator, Richard C. Shelton, MD, Vanderbilt University
Organization: Vanderbilt University Medical Center (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: RIS-BIP-4005; RIS-BIP-4005 (Other: Janssen Pharmaceutica)
Record Dates: First submitted 2007-12-11; First posted 2007-12-12 (Estimated); Results first posted 2017-07-31 (Actual); Last update posted 2017-07-31 (Actual); Status verified 2017-06

CONDITIONS: Bipolar Disorder
Keywords: Bipolar Disorder; Depression, Bipolar; Mania
MeSH Terms: conditions — Bipolar Disorder; Mania | interventions — Risperidone; Therapeutics

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Risperdal Consta (Experimental): Risperdal Consta injection in conjunction with existing treatment
  Interventions: Drug: Risperdal (risperidone) Consta
- Treatment As Usual (Active Comparator): Clinician and patient decide upon treatment, as in a non-research clinical setting. The only treatment exclusion is any form of risperidone.
  Interventions: Drug: Treatment as usual

INTERVENTIONS:
Drug: Risperdal (risperidone) Consta — Risperdal Consta (TM) will be administered every 2 weeks by deep intramuscular (IM) gluteal injection, by a trained health care professional. Injections will alternate between the two buttocks. The initial dose will be 25 mg IM every 2 weeks. A minimum dose of 25 mg. every 2 weeks will be maintained. At the clinician's discretion, the dose may be advanced to 37.5 mg. or 50 mg. In addition, the dose will be raised to 37.5 mg. or 50 mg. if the following conditions remain: (1) Young Mania Rating Scale (YMRS) score > 12; or (2) Evidence of impending relapse; and no dose limiting side effect. If the 25 mg. dose is not tolerated, the dose can be held temporarily; however, attempts will be made to achieve and maintain the dose at 25 mg. (or higher) until the end of the study period.
  Other Names: Risperidone long-acting injectible
  Arms: Risperdal Consta
Drug: Treatment as usual — Treatment was provided in this arm based solely on the choice of the treatment provider and participant. Treatment providers were not part of the study staff and were completely free to make treatment choices except that they were not allowed to select a long-acting injectible.
  Other Names: Usual care
  Arms: Treatment As Usual

SUMMARY:
This study will evaluate the relative effectiveness of risperidone Consta injections occurring every 2 weeks in contrast to treatment as usual in preventing symptomatic relapse and rates of rehospitalization or admission into respite care for bipolar patients.

Hypothesis: Risperdal Consta injections every 2 weeks will reduce the number of symptomatic relapses into mania, hypomania, mixed state, or depression, as shown by key indicators that include symptomatic relapse, rehospitalizations, emergency or urgent care visits, respite care, and intensive outpatient treatment as compared to treatment as usual.

DETAILED DESCRIPTION:
Bipolar disorder arguably represents the most difficult to treat of all psychiatric disorders. In fact, long-term stabilization is more the exception than the rule, and the majority of patients experience frequent relapses of illness. Studies have shown that both bipolar I and II patients spend about half of their weeks in a significant symptomatic state. Relapses and persistent illness result in substantial morbidity, mortality, and disability.

Symptomatic recurrences happen as a result of breakthrough symptoms during active treatment and intermittent non-adherence. Therefore, enhanced control of symptoms, coupled with ensured adherence, is very likely to improve the long-term outcome of this difficult-to-treat condition.

Risperidone has been shown to be effective in controlling symptoms of acute mania or mixed state in two registration monotherapy and one combination treatment study with lithium or valproate, as well as several smaller trials. However, longer-term treatment studies are relatively lacking. As well, although Risperdal Consta(TM) has been shown to be of benefit in prevention of relapse in patients with schizophrenia, relatively little longer-term data in bipolar disorder is available. Nonetheless, both risperidone and Risperdal Consta (TM) are likely to be highly efficacious for the maintenance prevention of relapse in bipolar disorder. Moreover, Risperdal Consta(TM) helps to ensure longer-term treatment effectiveness, both by better adherence and improved control of symptoms. The present study is intended to determine whether Risperdal Consta(TM) injections, added to ongoing pharmacotherapy, will improve outcome relative to treatment as usual.

ELIGIBILITY:
Inclusion Criteria:

* Be physically healthy
* 18-60 years of age
* Have a DSM-IV diagnosis of bipolar disorder in any phase, but without current psychotic features; with a history of symptomatic relapse on four or more occasions over the last year prior to the initiation of study for the treatment of bipolar disorder (type I or II, manic, hypomanic, mixed, or depressive type), with at least 1 in the previous 6 months.
* Have a screening Hamilton Rating Scale for Depression-17 item (HAM-D17) score of > 8 or a Young Mania Rating Scale (YMRS) > 8.

Exclusion Criteria:

* Have any medical condition that would preclude treatment with Risperdal Consta(TM)
* Have type 2 diabetes
* Have hyperlipidemia (baseline total cholesterol >280)
* Have any clinically significant unstable medical condition
* Have currently active psychotic symptoms (hallucinations or delusions) or carry a diagnosis of another psychotic disorder (schizophrenia, schizoaffective disorder, delusional disorder)
* Have a documentable history of non-response to Risperidal Consta (TM)
* Have a score of 4 on the suicide item (item 3) of the HAM-D scale and/or a determination by the investigator of significant suicide risk
* Require hospitalization between the screening and baseline visits, or require hospitalization immediately following baseline
* Have a medical contraindication or hypersensitivity to risperidone or Risperdal Consta (TM)

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 50 (Actual)
Dates: Start 2007-11; Primary Completion 2009-02 (Actual); Study Completion 2009-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Richard C Shelton, M.D., Principal Investigator — Vanderbilt University
Locations (1):
- Mental Health Cooperative, Inc., Nashville, Tennessee, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Referred by treating provider
Pre-assignment Details: Diagnostic review prior to randomization
Groups:
- Risperdal Consta: Risperdal Consta injection in conjunction with existing treatment
  Risperdal (risperidone) Consta: Risperdal Consta (TM) will be administered every 2 weeks by deep intramuscular gluteal injection, by a trained health care professional. Injections will alternate between the two buttocks. The initial dose will be 25 mg intramuscularly (IM) every 2 weeks. A minimum dose of 25 mg. every 2 weeks will be maintained. At the clinician's discretion, the dose may be advanced to 37.5 mg. or 50 mg. In addition, the dose will be raised to 37.5 mg. or 50 mg. if the following conditions remain: (1) Young Mania Rating Scale (YMRS) score > 12; or (2) Evidence of impending relapse; and no dose limiting side effect. If the 25 mg. dose is not tolerated, the dose can be held temporarily; however, attempts will be made to achieve and maintain the dose at 25 mg. (or higher) until the end of the study period.
Period: Overall Study
Arm/Group | Risperdal Consta | Treatment As Usual
Started | 25 | 25
Completed | 20 | 19
Not Completed | 5 | 6
Not completed — Lost to Follow-up | 3 | 6
Not completed — subject did not tolerate Consta | 1 | 0
Not completed — subject moved out of the area | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Risperdal Consta: Risperdal Consta injection in conjunction with existing treatment
  Risperdal (risperidone) Consta: Risperdal Consta (TM) will be administered every 2 weeks by deep intramuscular gluteal injection, by a trained health care professional. Injections will alternate between the two buttocks. The initial dose will be 25 mg IM every 2 weeks. A minimum dose of 25 mg. every 2 weeks will be maintained. At the clinician's discretion, the dose may be advanced to 37.5 mg. or 50 mg. In addition, the dose will be raised to 37.5 mg. or 50 mg. if the following conditions remain: (1) YMRS score > 12; or (2) Evidence of impending relapse; and no dose limiting side effect. If the 25 mg. dose is not tolerated, the dose can be held temporarily; however, attempts will be made to achieve and maintain the dose at 25 mg. (or higher) until the end of the study period.
- Total: Total of all reporting groups
Arm/Group | Risperdal Consta | Treatment As Usual | Total
Number analyzed (Participants) | 25 | 25 | 50
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 25 | 25 | 50
  >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: Years] | 42.8 (8.7) | 38.2 (10.2) | 40.5 (9.45)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 14 | 16 | 30
  Male | 11 | 9 | 20
Region of Enrollment [Number; unit: participants]
  United States | 25 | 25 | 50

OUTCOME MEASURES:

1. Primary Outcome: Number of Relapse-related Events Normalized to Unit Time
Description: The outcome was total number of events divided by number of months (normalized to unit time). This was be calculated by dividing the number of relapse related events by the number of months of participation. Relapse related events included: (1) YMRS score > 14 or MADRS > 15; (2) 20% or greater increase in the YMRS or MADRS scores from the previous study visit; (3) urgent care visit (psychiatric hospitalization; emergency department visit; referral for respite care, partial hospitalization, or intensive outpatient treatment) due to worsening mood symptoms; (4) a Clinical Global Impression Severity of Illness score >3; (5) syndromal relapse (Diagnostic and Statistical Manual of Mental Disorders, 4th Editionfor manic, hypomanic, major depressive, or mixed episode met); (6) withdrawal from the study due to inefficacy; and (7) necessary clinical medication adjustments (NCAs).
Time Frame: 12 months
Population: All randomized participants were analyzed.
Measure: Mean (Standard Deviation); unit: Events/month
Arm/Group | Risperdal Consta | Treatment As Usual
Number analyzed (Participants) | 25 | 25
Events/month | 5.34 (2.35) | 6.26 (3.24)

ADVERSE EVENTS:
Time Frame: 1 year
Description: Adverse effects spontaneously reported by participants.
Arm/Group | Risperdal Consta | Treatment As Usual
All-Cause Mortality (participants affected / at risk) | 0/25 | 0/25
Serious Adverse Events (participants affected / at risk) | 0/25 | 0/25
Other Adverse Events (participants affected / at risk) | 5/25 | 6/25
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Risperdal Consta (N=25) | Treatment As Usual (N=25)
Sedation (Nervous system disorders) | 3 (3) | 4 (4)
Weight gain (Metabolism and nutrition disorders) | 2 (2) | 3 (3)

LIMITATIONS AND CAVEATS:
This was not a blinded study.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No